CLINICAL TRIAL: NCT04744168
Title: Acupuncture Effect on the Rate of Maturation in Post Term Pregnancies.
Acronym: MATUPUNCTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDRCB 2020-A03023-36
Record Dates: First submitted 2021-01-22; First posted 2021-02-08 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Pregnancy Beyond 41 Week's Gestation
Keywords: Bishop's score; Maturation; Acupuncture; Pregnancy
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Women will be distributed randomly in the experimental or the placebo arm. They won't know that the point 16 HM isn't effective on cervix maturation. They will believe that both techniques work.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): In the experimental arm, pregnant women at term will benefit one or two acupuncture sessions with five points : 4GI, 6RP, 34VB,36E,3F. The first session at 41 amenorrhea weeks and the second at 41 amenorrhea weeks and 3 days if they are not delivered between the both.
  Interventions: Other: Acupuncture
- Placebo acupuncture (Placebo Comparator): In the placebo arm, pregnant women will benefit one or two acupuncture sessions with one point which is located outside the acupuncture meridian.
  The first session at 41 amenorrhea weeks and the second at 41 amenorrhea weeks and 3 days if they are not delivered between the both.
  Interventions: Other: Placebo Acupuncture

INTERVENTIONS:
Other: Acupuncture — Puncture of 5 points 4GI, 6RP, 34VB, 36E, 3F
  Arms: Acupuncture
Other: Placebo Acupuncture — Puncture of point HM
  Arms: Placebo acupuncture

SUMMARY:
Brief Summary Short description of the protocol intended for the lay public. Include a brief statement of the study hypothesis. (Limit: 5000 characters)

Example: The purpose of this study is to determine whether prednisone, methotrexate, and cyclophosphamide are effective in the treatment of rapidly progressive hearing loss in both ears due to autoimmune inner ear disease (AIED). The first purpose of this randomized study is to determine if five points of acupuncture : 4GI, 6RP, 34VB, 36E, 3F could improve the bishop score for prolonged pregnancies and decrease the rate of maturation.

The protocol of our study consists of proposing to the pregnant women one or two acupuncture sessions the term's day and three days later. Once the consent is signed, women are randomly included in the experimental or placebo arm. In the experimental arm, midwives puncture five points : 4GI, 6 RP, 34VB, 36E, 3F on each side while in the placebo arm, they puncture just one point : 16 HM on each side.

The maturation's rate between the two groups will be compared by a Fisher's exact test and analyzed in function parity (nulliparous or multiparous) and number of sessions (one or two) with a model of univariate and multivariate logistic regression.

DETAILED DESCRIPTION:
In maternity hospital center Corbeil-Essonnes, pregnant women have two monitoring consultations at term and three days later if they don't deliver between the two. At 41 weeks of amenorrhea and five days, women are convened in maternity for induction labour. Midwife determined Bishop's score with a vaginal exam to choose between a cervix's maturation (if bishop's score <5) or an induction of labour by oxytocin (if bishop's score>5).

The protocol of study consists of proposing to the pregnant women one or two acupuncture sessions the term's day and three days later. Once the consent is signed, women are randomly included in the experimental or placebo arm. In the experimental arm, midwives puncture five points : 4GI, 6 RP, 34VB, 36E, 3F on each side while in the placebo arm, they puncture just one point : 16 HM on each side.

At each consultation, the midwife collects the bishop's score to compare the average of it between the two arms and evaluate the rate of maturation.

The maturation's rate between the two groups will be compared by a Fisher's exact test and analyzed in function parity (nulliparous or multiparous) and number of sessions (one or two) with a model of univariate and multivariate logistic regression.

Finally, the average duration of induction labour will analyze, duration of labour and delivery route between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous or multipares with physiological pregnancy at 41 weeks
* Cephalic foetal presentation,
* Healthy or unicicatricial uterus,
* Major patientes,
* Speaking french,
* Term of the pregnancy determinated with a dating ultrasound between 11 weeks and 13 weeks+ 6 days,
* Having signed the form of consent participation.

Exclusion Criteria:

* Foetal or maternal diseases requiring a maturation before 41 weeks : pre eclampsia, pre-existing diabetes, imbalance gestational diabetes, threat premature delivery treat with tocolytic, macrosomia or intrauterine growth retardation,
* Diseases discoveries at 41 weeks : pre eclampsia, moves of the baby decrease, low amniotic fluid,anomalies of the foetal heartbeat
* Circled pregnancy,
* Twins or more,
* Foetal death in utero, medical termination of pregnancy,
* Unstuck membranes,
* Minor patients
* Patients who benefited acupuncture during pregnancy ,
* Imprecise term of delivery,
* Podalic presentation
* Patients under supervision or curatorship,
* Patients without social security.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Bishop score | At 41 weeks of amenorrhea
  cervix score is a pre-labor scoring system to assist in predicting whether induction of labor will be required (The highest possible score is 13 and the lowest possible score is 0)
Bishop score | 3 days after the term of pregnancy
  cervix score is a pre-labor scoring system to assist in predicting whether induction of labor will be required
Bishop score | 5 days after the term of pregnancy
  cervix score is a pre-labor scoring system to assist in predicting whether induction of labor will be required

SECONDARY OUTCOMES:
Rate spontaneous labour | At 41 weeks 5 days of amenorrhea
  comparison of spontaneous labour's number in the two groups between 41 weeks of amenorrhea and 41 weeks of amenorrhea and five days.
Duration labor | At 41 weeks 5 days of amenorrhea
  comparison of average number of hours between entry into the delivery room and the delivery, in the two groups.
Rate of delivery with medical intervention | At 41 weeks 5 days of amenorrhea
  comparison medical intervention's number in the two groups.
Rate of delivery by cesarean | At 41 weeks 5 days of amenorrhea
  comparison cesarean's number in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No